CLINICAL TRIAL: NCT02980978
Title: diEtitiaNs Helping pAtieNts CarE for Diabetes (ENHANCED)
Acronym: ENHANCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ENHANCED
Record Dates: First submitted 2016-11-15; First posted 2016-12-02 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Individuals assigned to the intervention group will have supplemental care provided by a registered dietitian/certified diabetes educator which includes counseling on lifestyle to improve diabetes and overall health. Additionally, individuals in this group may be started on medications (or adjustments to current medications) for blood pressure, cholesterol or blood glucose to meet diabetes care goals
  Interventions: Behavioral: Coaching
- Standard of Care (No Intervention): Individuals will be followed by their Primary Care Provider as standard of care and per usual clinical need

INTERVENTIONS:
Behavioral: Coaching — Focus on nutrition, activity and appropriate medication use and adherence
  Arms: Intervention

SUMMARY:
This study aims to randomly assign individuals with type 2 diabetes into the ENHANCED randomized control trial. The study is being conducted by the Minneapolis Heart Institute Foundation (MHIF) and will have two study sites 1) Hutchinson Health and 2) New Ulm Medical Center. The study is primarily funded through the Academy of Nutrition and Dietetics (AND).

The study will examine the impact of a registered dietitian-led, primary care integrated, telemedicine program on diabetes care measures (the 'D5') over one year as compared to usual care. The D5 goals include: blood pressure <140/90 mmHg, taking a statin as appropriate, A1c <8%, not using tobacco and taking an aspirin as appropriate.

DETAILED DESCRIPTION:
Individuals will be invited to attend a baseline visit where they will have lab work done, anthropometrics (height, weight, waist circumference) and complete a lifestyle assessment. They will formally consent to participation by signing a study consent form. The same measures will be collected after completion of the one year study.

Study participants will receive two sessions of free lab work, a diabetes education book, and brief coaching with a registered dietitian/certified diabetes educator. In addition, those randomized to the phone coaching will have access to a registered dietitian/certified diabetes educator on a monthly basis for one year of personalized health coaching for free. The intent of this coaching is to help individuals achieve diabetes "optimal" care or meeting all 5 Diabetes Care measures (blood glucose, blood pressure, tobacco use, statin and aspirin use).

This program is designed to complement usual clinic-based primary care, with coaches documenting lab, biometrics and medication adjustments in the EHR, along with documenting phone encounters and communicating directly with patients' PCPs as needed. Documentation in the EHR uses an order created specifically for the study indicating the patient's research status.

Lab work required as part of this research study at baseline and 12 months is covered by the study. Any lab work and/or medication co-pays or fees outside of the baseline and 12 month study visits are the responsibility of the patient and/or their insurance

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 2 Diabetes
2. Individuals who are not meeting 3 or more D5 goals,
3. Have had a visit with a provider within the last 2 years

Exclusion Criteria:

1. Type 1 Diabetes
2. Chronic kidney disease (GFR <30)
3. HIV
4. Institutional residence
5. Major cognitive or language barrier (as determined by program enrollment staff)
6. Other active end-stage disease (e.g., late stage cancer or pulmonary disease)
7. Actively receiving cancer treatment
8. Pregnant

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miedema, MD, Principal Investigator — Minneapolis Heart Institute Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benson GA, Sidebottom A, Hayes J, Miedema MD, Boucher J, Vacquier M, Sillah A, Gamam S, VanWormer JJ. Impact of ENHANCED (diEtitiaNs Helping pAtieNts CarE for Diabetes) Telemedicine Randomized Controlled Trial on Diabetes Optimal Care Outcomes in Patients with Type 2 Diabetes. J Acad Nutr Diet. 2019 Apr;119(4):585-598. doi: 10.1016/j.jand.2018.11.013. Epub 2019 Jan 31. PMID 30711463

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Standard of Care
Started | 60 | 58
Completed | 54 | 50
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard of Care | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 50 | 98
  >=65 years | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (10.2) | 60.0 (8.66) | 59.9 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 32 | 33 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 56 | 52 | 108
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 60 | 58 | 118

OUTCOME MEASURES:

1. Primary Outcome: A1c (Laboratory Assessment)
Description: The count of participants represents the number of individuals meeting A1c less than 8% at follow up
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 54 | 50
Participants | 35 | 35

2. Other Pre Specified Outcome: Blood Pressure (Calibrated Cuff Measurement- Average of 3 Readings)
Description: The count of participants represents the number of individuals meeting blood pressure less than 140/90 at follow up
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 54 | 50
Participants | 24 | 20

3. Other Pre Specified Outcome: Tobacco Use (Self-reported Questionnaire)
Description: The count of participants represents those not using tobacco at follow up
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 54 | 50
Participants | 44 | 40

4. Other Pre Specified Outcome: Statin Use (as Noted in EMR)
Description: The count of participants represents those taking a statin as indicated at follow up
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 54 | 50
Participants | 50 | 32

5. Other Pre Specified Outcome: Aspirin Use (as Noted in EMR)
Description: The count of participants represents taking aspirin as indicated at follow up
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 54 | 50
Participants | 45 | 34

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT02980978/Prot_SAP_000.pdf